CLINICAL TRIAL: NCT05581485
Title: Comparison of Dexmedetomidine and Superior Laryngeal Nerve Block for Non-Intubated Endoscopic Laryngeal Surgery With Spontaneous Breathing Using Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): A Randomized Controlled Trial
Brief Title: Dex vs SLNB in Spontaneous Breathing Via THRIVE for Laryngeal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Yuan-Yi Chia, Chief of Anesthesiology, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSVGH22-CT8-38
Record Dates: First submitted 2022-10-04; First posted 2022-10-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Endoscopic Laryngeal Surgery
Keywords: Laryngomicrosurgery; Nonintubation; spontaneous breathing; dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine Infusion Arm for Non-Intubated Laryngeal Surgery Using THRIVE (Experimental): This arm involves patients undergoing endoscopic laryngeal surgery under non-intubated general anesthesia with spontaneous breathing, supported by transnasal humidified rapid-insufflation ventilatory exchange (THRIVE). Patients receive an intravenous loading dose of dexmedetomidine (1 µg/kg over 10 minutes), followed by a continuous infusion (1 µg/kg/h) for sedation and analgesia. No regional nerve blocks are performed in this arm. Supplemental propofol is titrated via target-controlled infusion (TCI) to maintain BIS levels between 40-60. Topical 10% lidocaine is applied to the airway before insertion of the laryngoscope. Intraoperative fentanyl may be given as needed based on hemodynamic responses.
  Interventions: Drug: Dexmetedomedine infusion
- Superior Laryngeal Nerve Block (SLNB) (Active Comparator): This arm includes patients undergoing non-intubated endoscopic laryngeal surgery with spontaneous breathing, supported by transnasal humidified rapid-insufflation ventilatory exchange (THRIVE). After induction with propofol (via TCI) and standard premedication, bilateral ultrasound-guided superior laryngeal nerve blocks are performed using 5 mL of 1% lidocaine on each side for regional analgesia. No dexmedetomidine is administered in this group. Anesthesia is maintained with propofol titrated to a BIS range of 40-60. Additional fentanyl may be administered intraoperatively as needed to control sympathetic responses. Topical 10% lidocaine is applied to the airway prior to laryngoscope insertion.
  Interventions: Procedure: Ultrasound-Guided Superior Laryngeal Nerve Block (SLNB)

INTERVENTIONS:
Drug: Dexmetedomedine infusion — Patients received a loading dose of dexmedetomidine at 1 µg/kg over 10 minutes, followed by a continuous infusion at 1 µg/kg/h throughout the procedure. This regimen was combined with TIVA (propofol) and THRIVE to support spontaneous breathing during endoscopic laryngeal surgery.
  Arms: Dexmedetomidine Infusion Arm for Non-Intubated Laryngeal Surgery Using THRIVE
Procedure: Ultrasound-Guided Superior Laryngeal Nerve Block (SLNB) — Following anesthesia induction, patients received bilateral ultrasound-guided superior laryngeal nerve blocks using 5 mL of 1% lidocaine per side. This intervention was combined with total intravenous anesthesia (TIVA) using propofol and high-flow nasal oxygenation (THRIVE) to maintain spontaneous respiration during endoscopic laryngeal surgery.
  Arms: Superior Laryngeal Nerve Block (SLNB)

SUMMARY:
This prospective, randomized controlled trial evaluated the efficacy and safety of two anesthetic strategies-dexmedetomidine infusion and ultrasound-guided superior laryngeal nerve block (SLNB)-in patients undergoing non-intubated endoscopic laryngeal surgery under spontaneous breathing supported by Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE). The primary outcome was the arterial partial pressure of carbon dioxide (PaCO₂), measured at three time points: before oxygenation, at the end of surgery, and in the post-anesthesia care unit (PACU). Secondary outcomes included other arterial blood gas parameters, hemodynamic variables, and surgeon satisfaction scores.

DETAILED DESCRIPTION:
Detailed Description:

This prospective, single-center randomized controlled trial was conducted to compare two anesthetic strategies-Dexmedetomidine infusion and ultrasound-guided bilateral superior laryngeal nerve block (SLNB)-for non-intubated endoscopic laryngeal surgery performed under spontaneous respiration with high-flow nasal oxygenation (THRIVE). The study was carried out at Kaohsiung Veterans General Hospital, Taiwan.

Patients aged 20 to 80 years scheduled for elective microlaryngeal surgery were enrolled and randomly assigned to either the Dexmedetomidine (Dex) group or the SLNB group. Both groups received total intravenous anesthesia (TIVA) with propofol and oxygenation via transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) to facilitate tubeless anesthesia. The Dex group received a loading dose of Dexmedetomidine (1 µg/kg over 10 minutes) followed by continuous infusion (1 µg/kg/h), while the SLNB group underwent bilateral ultrasound-guided nerve blocks with 1% lidocaine.

The primary outcome was the arterial partial pressure of carbon dioxide (PaCO₂) measured at three time points: before oxygenation (baseline), at the end of surgery, and 15 minutes after arrival in the post-anesthesia care unit (PACU). Secondary outcomes included arterial blood gas parameters (PaO₂, pH), intraoperative hemodynamic variables (HR, SBP, DBP, MAP), and surgeon satisfaction scores.

The goal of this study was to evaluate whether Dexmedetomidine, which offers both sedative and analgesic properties while preserving spontaneous breathing, could serve as a viable alternative to regional nerve block in the context of shared-airway surgery. Particular attention was given to the risk of carbon dioxide accumulation and respiratory acidosis associated with Dexmedetomidine.

This trial provides important insights into the safety and efficacy of two distinct anesthetic modalities for performing non-intubated endoscopic laryngeal surgery and contributes to the ongoing optimization of airway management strategies in tubeless anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are between 20-80 years old.
* Patients undergoing endoscopic laryngeal surgery.
* Anesthesiologists rated ASA as between I and III.

Exclusion Criteria:

* Having drug dependence and drinking habits.
* Abnormal heart, liver and kidney function.
* Allergic reactions to narcotic drugs.
* Emergency surgery.
* pregnancy.
* Refuse to participate.
* BMI ≥ 35 kg/m2.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Perioperative PaCO2 | From pre-induction through 15 minutes postoperatively
  Arterial blood gas was collected and analyzed at three time points to assess changes in PaCO₂ as the primary outcome:
  1. At baseline (after preoxygenation, prior to induction)
  2. Immediately after completion of endoscopic laryngeal surgery
  3. Fifteen minutes after arrival in the post-anesthesia care unit (PACU)

SECONDARY OUTCOMES:
Arterial Oxygenation (PaO₂) | From pre-induction through 15 minutes postoperatively
  Arterial partial pressure of oxygen (PaO₂) measured via ABG at three time points: preoxygenation baseline, immediately post-surgery, and 15 minutes after PACU arrival.
Mean Arterial Pressure (MAP) | Preoperative, intraoperative (every 5 minutes), and 15 minutes postoperatively in the PACU
  Monitoring of mean arterial pressure at defined intervals to evaluate cardiovascular responses to anesthetic strategy.
Heart rate | Preoperative, intraoperative (every 5 minutes), and 15 minutes postoperatively in the PACU
  Assessment of heart rate variability across the surgical timeline to monitor hemodynamic stability.
Surgeon stress score | Immediately after completion of the surgical procedure
  Subjective evaluation of the surgeon's intraoperative stress level, based on surgical field visibility, patient movement, and anesthetic stability. The score is rated on a 6-point scale from 0 to 5, where:
  0 = No stress
  1. = Minimal stress
  2. = Mild stress
  3. = Moderate stress
  4. = High stress
  5. = Extremely high stress
Arterial pH | Baseline, end of surgery, PACU (15 minutes post-arrival)
  Arterial pH will be measured at three time points:
  1. preoxygenation (baseline),
  2. immediately after the end of endoscopic laryngeal surgery,
  3. 15 minutes after arrival in the post-anesthesia care unit (PACU).

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wei Hsieh, physician, Study Director — Kaohsiung Veterans General Hospital.; Ting Shou Chang, physician, Study Director — Kaohsiung Veterans General Hospital.; Chih Chi Tsai, RA, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan, Taiwan

REFERENCES:
- [Background] Yang SH, Wu CY, Tseng WH, Cherng WY, Hsiao TY, Cheng YJ, Chan KC. Nonintubated laryngomicrosurgery with Transnasal Humidified Rapid-Insufflation Ventilatory Exchange: A case series. J Formos Med Assoc. 2019 Jul;118(7):1138-1143. doi: 10.1016/j.jfma.2018.11.009. Epub 2018 Dec 3. PMID 30522856
- [Background] Gustafsson IM, Lodenius A, Tunelli J, Ullman J, Jonsson Fagerlund M. Apnoeic oxygenation in adults under general anaesthesia using Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) - a physiological study. Br J Anaesth. 2017 Apr 1;118(4):610-617. doi: 10.1093/bja/aex036. PMID 28403407
- [Background] W.Abd El Megid, W., & Nassar, A. M. (2009). The analgesic and sedative properties of dexmedetomidine infusion after uvulopalatopharyngoplasty. The Egyptian Journal of Hospital Medicine, 36(1), 421-433.
- [Background] Gemechu BM, Gebremedhn EG, Melkie TB. Risk factors for postoperative throat pain after general anaesthesia with endotracheal intubation at the University of Gondar Teaching Hospital, Northwest Ethiopia, 2014. Pan Afr Med J. 2017 Jun 16;27:127. doi: 10.11604/pamj.2017.27.127.10566. eCollection 2017. PMID 28904657
- [Background] Ahmed A, Saad D, Youness AR. Superior laryngeal nerve block as an adjuvant to General Anesthesia during endoscopic laryngeal surgeries. Egyptian Journal of Anaesthesia 2015;31:167-74.
- [Background] Naaz S, Ozair E. Dexmedetomidine in current anaesthesia practice- a review. J Clin Diagn Res. 2014 Oct;8(10):GE01-4. doi: 10.7860/JCDR/2014/9624.4946. Epub 2014 Oct 20. PMID 25478365
- [Background] Abdelmageed WM, Elquesny KM, Shabana RI, Abushama HM, Nassar AM. Analgesic properties of a dexmedetomidine infusion after uvulopalatopharyngoplasty in patients with obstructive sleep apnea. Saudi J Anaesth. 2011 Apr;5(2):150-6. doi: 10.4103/1658-354X.82782. PMID 21804794 (Retraction: PMID 31998047 Saudi J Anaesth. 2020 Jan-Mar;14(1):144)
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Background] Booth AWG, Vidhani K, Lee PK, Thomsett CM. SponTaneous Respiration using IntraVEnous anaesthesia and Hi-flow nasal oxygen (STRIVE Hi) maintains oxygenation and airway patency during management of the obstructed airway: an observational study. Br J Anaesth. 2017 Mar 1;118(3):444-451. doi: 10.1093/bja/aew468. PMID 28203745